CLINICAL TRIAL: NCT04383808
Title: Clinical Translation of a Novel Brain PET Insert for Simultaneous PET/MR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Craig Levin, Professor, Radiology/ Nuclear Medicine, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-55044
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Brain Disease
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Arm-1 (Experimental): 20 participants will be recruited, inject with radiopharmaceutical, and imaged on the 3T PETMR with PET insert.
  Interventions: Diagnostic Test: Injected radiotracer with PET Insert
- Arm-2 (Experimental): 20 participants will be recruited from other imaging studies that have been already injected (pre-injected) with a radiopharmaceutical. These subjects wont receive an additional injection of radiopharmaceutical.
  Interventions: Diagnostic Test: Pre-injected group with PET insert

INTERVENTIONS:
Diagnostic Test: Injected radiotracer with PET Insert — 1. Informed consent will be obtained before beginning any study procedures.
  2. Participants will receive a small quantity of an FDA approved radiotracer. The PET insert is placed within a 3T MRI scanner, where PET and MRI imaging will be completed.
  Arms: Arm-1
Diagnostic Test: Pre-injected group with PET insert — 1. Informed consent will be obtained before beginning any study procedures.
  2. Participants who have received radiotracer for another PET imaging system. The PET insert is placed within a 3T MRI scanner, where PET and MRI imaging will be completed.
  Arms: Arm-2

SUMMARY:
The primary goal of this project is to study the feasibility of a brain-dedicated PET insert for an MR scanner for simultaneous acquisition of PET/MR images of human brains. The study will also allow us to compare the imaging performance of the investigator's brain-dedicated PET insert against a commercial whole-body permanently integrated PET/MRI system using a common radiopharmaceutical.

DETAILED DESCRIPTION:
This study will enroll up to 40 participants.

1. 20 participants at Stanford injected with an FDA-approved PET tracer (e.g. amyloid, FDG, etc.), and
2. 20 participants from Stanford who have been pre-injected with a radiopharmaceutical for a study on another PET imaging system

ELIGIBILITY:
Inclusion Criteria:

1. Whole body radiation dose within the last year of less than 5000 mrem
2. Subjects intended for injected tracer studies (not associated with another study) must be willing/able to undergo injection of 6-12 mCi of either FDG or Neuraceq radiotracer. Both tracers are FDA approved
3. Subjects will be at least 21 years of age
4. Subject provides written informed consent
5. Subject is deemed healthy by the PI by via self-reported questionnaire

Exclusion Criteria:

1. For patients who will be receiving a tracer injection, no known allergy to the imaging agents
2. Participant has a history of or current diagnosis of cancer
3. Participant is pregnant or nursing
4. Metallic implants (contraindicated for MRI)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
PETMR image | Up to 24 months
  The key specific measurement is the resulting PET/MR image obtained from the single subject scan.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States